CLINICAL TRIAL: NCT01621347
Title: Retrospective Study: Evaluation of Antiretroviral Adherence During Pregnancy and Postpartum Using Electronic Monitoring Data
Brief Title: Antiretroviral Adherence Evaluation in HIV Pregnant and Postpartum Women
Status: Completed | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Swiss HIV Cohort Study (Network)
Responsible Party: Principal Investigator, Marie Schneider, Pharmacist, PhD, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Other Study IDs: 48/12
Record Dates: First submitted 2012-05-31; First posted 2012-06-18 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infection; Pregnancy
Keywords: HIV; Pregnancy; Postpartum; Women; Medication Adherence
MeSH Terms: conditions — HIV Infections; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare adherence to antiretroviral therapy during pregnancy and postpartum, and to record adherence barriers and facilitators.

DETAILED DESCRIPTION:
Data of all consecutive pregnant women included in the adherence enhancing program of the Pharmacy, Department of ambulatory care & community medicine, are collected. In this program, adherence is measured and enhanced by electronic monitoring, pill count, motivational interviewing and interdisciplinary collaboration. Electronic monitoring data are collected during pregnancy and postpartum, and compared. Barriers and facilitators are collected using interview's marks.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women
* HIV-positive
* Antiretroviral medication delivered in electronical monitors

Exclusion Criteria:

* Monitored period during pregnancy < 1 month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant and Postpartum Women enrolledin the HIV adherence program at the pharmacy of Department of Ambulatory Care and Community Medicine in Lausanne
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in patient adherence during pregnancy and postpartum | before delivery (1 to 9 month) and postpartum (6 month)
  By electronic drug monitoring, pill count and subject interviews' marks

SECONDARY OUTCOMES:
Adherence barriers and facilitators | pregnancy and postpartum (6 months)
  Data recorded in subject's interview marks

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Paule Schneider, PhD, Study Chair — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Aurélie Gertsch, PhD-Student, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Olivier Bugnon, Professor, Study Chair — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Odile Michel, Student, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Matthias Cavassini, M.D, Study Chair — Centre Hosppitalier Universitaire Vaudois
Locations (1):
- Policlinique Médicale Universitaire, Lausanne, Canton of Vaud, Switzerland